CLINICAL TRIAL: NCT05442125
Title: Whether Using DNA Methylome to Select Embryos Can Increase the Live Birth Rate During Assisted Reproductive Technology: A Multicenter, Randomized , Open-label Clinical Trial.
Brief Title: First Live Birth Rate With eSET After Preimplantation Methylome Screening (PIMS) Versus Conventional In-vitro Fertilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: RenJi Hospital (Other); Reproductive & Genetic Hospital of CITIC-Xiangya (Other); Nanjing Maternity and Child Health Care Hospital (Other); ShangHai Ji Ai Genetics & IVF Institute (Other); Suzhou Municipal Hospital (Other); The First Hospital of Jilin University (Other); Sir Run Run Shaw Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The Second Hospital of Hebei Medical University (Other); Third Affiliated Hospital of Zhengzhou University (Other); Ruijin Hospital (Other); International Peace Maternity and Child Health Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Hainan Medical University (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Fujian Maternity and Child Health Hospital (Other); General Hospital of Ningxia Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); 900 Hospital of Joint Logistics Support Force of PLA (Other); Guangzhou Womenand Children's Medical Center (Unknown); Changhai Hospital (Other); Shenzhen Maternity & Child Healthcare Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Liuzhou Hospital of Guangzhou Women and Children's Medical Center (Unknown); Jining Medical University (Other); Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Academician, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIMS-IVF
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Reproductive Techniques, Assisted; DNA Methylation
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMS group (Experimental): Couples in the PIMS group will have up to 6 blastocysts screened with PIMS and a single euploid embryo with the optimal state of whole-genome DNA methylation and the highest morphologic score will be selected for the initial transfer. The optimal state of whole-genome DNA methylation includes methylation level closest to the optimal level (0.26 according to our preliminary results) and proper methylation state for some specific regions.
  Interventions: Other: Using DNA methylome to select embryos
- Conventional-IVF group (Active Comparator): For women between 20 and 37 years of age,couples in the conventional-IVF group will have a single best blastocyst by morphologic criteria selected for the initial transfer.For women over 37 years old, couples in the PGT-A group will have up to 6 blastocysts tested with PGT-A and a single euploid embryo with the highest morphologic score will be selected for the initial transfer.
  Interventions: Other: Using morphologic score to select embryos

INTERVENTIONS:
Other: Using DNA methylome to select embryos — DNA methylation level Embryo with methylation level closest to the optimal level (from one couple patients) is the one for embryonic transfer to uterus
  Arms: PIMS group
Other: Using morphologic score to select embryos — blastocyst will transferred according to morphologic score or blastocysts will be biopsied on trophectoderm, sequenced with next-generation sequencing (NGS). Euploidy will transferred one by one according to morphologic score.
  Arms: Conventional-IVF group

SUMMARY:
To determine whether using DNA methylome to select embryos can increase the live birth rate.

DETAILED DESCRIPTION:
The rationale for the study is to establish the risk/benefit ratio of PIMS in women with in vitro fertilization (IVF) treatment, as DNA methylome is a potential biomarker in blastocyst selection in assited reproductive technology (ART). DNA methylation plays an important role during embryogenesis, global abnormal methylome reprogramming often occurs in human embryos, and DNA methylome pattern is associated with live birth rate. However, there is still no technology using DNA methylome as an indicator in preimplantation embryo screening. Recent paper reported that using Pre-implantation Methylome Screening (PIMS) can select embryos with better methylation state and euploid chromosomes. The efficiency of PIMS needs further validation through randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women who plan to undergo IVF/ICSI/PGT-A treatment.
2. Women aged 20 years and older.

b) Women who obtain 2 or more good-quality blastocysts that defined as morphological score of inner cell mass B or A, trophectoderm C or better, and grade 4 or better on Day 5 of embryo culture.

Exclusion Criteria:

4.2 Exclusion Criteria

1. Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus unicornate, bicornate, or duplex); untreated uterine septum, submucous myoma, or endometrial polyp(s); or with history of intrauterine adhesions.
2. Women who are indicated and planned to undergo preimplantation genetic testing for structural rearrangements (PGT-SR) or preimplantation genetic testing for monogenic (PGT-M).
3. Women who use donated oocytes or sperm to achieve pregnancy;
4. Women with contraindication for assisted reproductive technology or for pregnancy, such as poorly controlled Type I or Type II diabetes; undiagnosed liver disease or dysfunction (based on serum liver enzyme testing); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; uncontrolled hypertension, known symptomatic heart disease; history of or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma; undiagnosed vaginal bleeding.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1146 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
live birth rate of initial embryo transfer | 22 months
  Live birth rate is defined as delivery of any viable infant at 28 weeks or more of gestation, after initial embryo transfer in women using the embryos selected through PIMS or PGT-A or morphological criteria alone.

SECONDARY OUTCOMES:
Good Birth Outcome rate | 36 months
  Defined as a live birth of an infant born at ≥ 37 weeks, with a birth weigh between 2500 and 4000g and without a major congenital anomaly
Clinical pregnancy rate | 36 months
  Twenty days after conception, transvaginal ultrasonography will be performed. Clinical pregnancy will be diagnosed with detection of an intrauterine gestational sac.
Pregnancy loss rate | 36 months
  Number of pregnancy losses / number of clinical pregnancies after transfer.
Multiple pregnancy rate | 36 months
  Number of multiple pregnancy/number of clinical pregnancies after transfer.
Duration of pregnancy | 36 months
  Duration of pregnancy is the period between conception and birth.
Birth weight | 36 months
  Weight of newborns at delivery.
Maternal complications | 48 months
  Number of pregnancies with complications / number of pregnancies.
Neonatal complications | 48 months
  Number of live births with neonatal complications / number of live births.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Gao, Professor, Study Director — Center for Reproductive Medicine, Shandong University; Yun Sun, Professor, Principal Investigator — Center for Reproductive Medicine, Ren Ji Hospital, School of Medicine,Shanghai Jiao Tong University; Ge Lin, Professor, Principal Investigator — Clinical Research Center for Reproduction and Genetics in Hunan Province, Reproductive and Genetic Hospital of CITIC-XIANGYA; Xiufeng Ling, Professor, Principal Investigator — Department of Reproductive Medicine, Women's Hospital of Nanjing Medical University, Nanjing Maternity and Child Health Care Hospital; Xiaoxi Sun, Professor, Principal Investigator — Shanghai Ji Ai Genetics and IVF Institute, Obstetrics and Gynecology Hospital, Fudan University; Hong Li, Professor, Principal Investigator — Center for reproduction and genetics,suzhou municipal hospital; Ruizhi Liu, Professor, Principal Investigator — Center for Reproductive Medicine, Center for Prenatal Diagnosis First Hospital, Jilin University; Songying Zhang, Professor, Principal Investigator — Assisted Reproduction Unit, Sir Run Run Shaw Hospital, Zhejiang University School of Medicine; Shuyun Zhao, Professor, Principal Investigator — Center for Reproductive Medicine, The Affiliated Hospital of Guizhou Medical University; Guimin Hao, Professor, Principal Investigator — The Second Hospital of Hebei Medical University; Yichun Guan, Professor, Principal Investigator — Department of Reproductive Medicine, the Third Affiliated Hospital of Zhengzhou University; Aijun Zhang, Professor, Principal Investigator — Reproductive Medical Center of Ruijin Hospital, School of Medicine,Shanghai Jiao Tong University; Wen Li, Professor, Principal Investigator — International Peace Maternity and Child Health Hospital, School of Medicine, Shanghai Jiao Tong University; Cuilian Zhang, Professor, Principal Investigator — Reproductive Medical Center, Henan Provincial People's Hospital; Yanlin Ma, Professor, Principal Investigator — The First Affiliated Hospital of Hainan Medical University; Yunxia Cao, Professor, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Beihong Zhen, Professor, Principal Investigator — Fujian Maternity and Child Health Hospital College of Clinical Medicine for Obstetrics & Gynecology and Pediatrics, Fujian Medical University; Junli Zhao, Professor, Principal Investigator — The General Hospital of Ningxia Medical University; Xiang Ma, Professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Yun Liu, Professor, Principal Investigator — 900 Hospital of Joint Logistics Support Force of PLA; Ling Sun, Professor, Principal Investigator — Guangzhou Womenand Children's Medical Center; Hongli Yan, Professor, Principal Investigator — Changhai Hospital; Xuemei Li, Professor, Principal Investigator — Shenzhen Maternity & Child Healthcare Hospital; Haitao Zeng, Professor, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University; Li Fan, Professor, Principal Investigator — Liuzhou Hospital of Guangzhou Women and Children's Medical Center; Aijun Yang, Professor, Principal Investigator — Jining Medical University; Isarin Thanaboonyawat, Doctor, Principal Investigator — Siriraj Hospital
Locations (28):
- China (27):
  - Shandong University, Jinan, Shandong
  - Center for Reproductive Medicine, Center for Prenatal Diagnosis First Hospital, Jilin University, Changchun
  - Clinical Research Center for Reproduction and Genetics in Hunan Province, Reproductive and Genetic Hospital of CITIC-XIANGYA, Changsha
  - 900 th Hospital of Joint Logistics Support Force, Fuzhou
  - Fujian Maternity and Child Health Hospital College of Clinical Medicine for Obstetrics & Gynecology and Pediatrics, Fujian Medical University, Fuzhou
  - Guangzhou Womenand Children's Medical Center, Guanzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guanzhou
  - Center for Reproductive Medicine, The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The first affiliated hospital of Hainan Medical University, Haikou
  - Assisted Reproduction Unit, Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Center for Reproductive Medicine, Shandong University, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Liuzhou Hospital of Guangzhou Women and Children's Medical Center, Liuchow
  - Department of Reproductive Medicine, Women's Hospital of Nanjing Medical University, Nanjing Maternity and Child Health Care Hospital, Nanjing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Center for Reproductive Medicine, Ren Ji Hospital, School of Medicine,Shanghai Jiao Tong University, Shanghai
  - Changhai Hospital, Shanghai
  - International Peace Maternity and Child Health Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Reproductive Medical Center of Ruijin Hospital, School of Medicine,Shanghai Jiao Tong University, Shanghai
  - Shanghai Ji Ai Genetics and IVF Institute, Obstetrics and Gynecology Hospital, Fudan University, Shanghai
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Center for reproduction and genetics,suzhou municipal hospital, Suzhou
  - The General Hospital of Ningxia Medical University, Yinchuan
  - Department of Reproductive Medicine, the Third Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Reproductive Medical Center, Henan Provincial People's Hospital, Zhengzhou
- Siriraj hospital, Mahidol university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brezina PR, Kutteh WH. Clinical applications of preimplantation genetic testing. BMJ. 2015 Feb 19;350:g7611. doi: 10.1136/bmj.g7611. PMID 25697663
- [Result] Hassold T, Chen N, Funkhouser J, Jooss T, Manuel B, Matsuura J, Matsuyama A, Wilson C, Yamane JA, Jacobs PA. A cytogenetic study of 1000 spontaneous abortions. Ann Hum Genet. 1980 Oct;44(2):151-78. doi: 10.1111/j.1469-1809.1980.tb00955.x. PMID 7316468
- [Result] Dahdouh EM, Balayla J, Audibert F; Genetics Committee; Wilson RD, Audibert F, Brock JA, Campagnolo C, Carroll J, Chong K, Gagnon A, Johnson JA, MacDonald W, Okun N, Pastuck M, Vallee-Pouliot K. RETIRED: Technical Update: Preimplantation Genetic Diagnosis and Screening. J Obstet Gynaecol Can. 2015 May;37(5):451-63. doi: 10.1016/s1701-2163(15)30261-9. PMID 26168107
- [Result] Kalousek DK, Pantzar T, Tsai M, Paradice B. Early spontaneous abortion: morphologic and karyotypic findings in 3,912 cases. Birth Defects Orig Artic Ser. 1993;29(1):53-61. No abstract available. PMID 8280893
- [Result] Rubio C, Bellver J, Rodrigo L, Castillon G, Guillen A, Vidal C, Giles J, Ferrando M, Cabanillas S, Remohi J, Pellicer A, Simon C. In vitro fertilization with preimplantation genetic diagnosis for aneuploidies in advanced maternal age: a randomized, controlled study. Fertil Steril. 2017 May;107(5):1122-1129. doi: 10.1016/j.fertnstert.2017.03.011. Epub 2017 Apr 19. PMID 28433371
- [Result] Sacchi L, Albani E, Cesana A, Smeraldi A, Parini V, Fabiani M, Poli M, Capalbo A, Levi-Setti PE. Preimplantation Genetic Testing for Aneuploidy Improves Clinical, Gestational, and Neonatal Outcomes in Advanced Maternal Age Patients Without Compromising Cumulative Live-Birth Rate. J Assist Reprod Genet. 2019 Dec;36(12):2493-2504. doi: 10.1007/s10815-019-01609-4. Epub 2019 Nov 12. PMID 31713776
- [Result] Yan J, Qin Y, Zhao H, Sun Y, Gong F, Li R, Sun X, Ling X, Li H, Hao C, Tan J, Yang J, Zhu Y, Liu F, Chen D, Wei D, Lu J, Ni T, Zhou W, Wu K, Gao Y, Shi Y, Lu Y, Zhang T, Wu W, Ma X, Ma H, Fu J, Zhang J, Meng Q, Zhang H, Legro RS, Chen ZJ. Live Birth with or without Preimplantation Genetic Testing for Aneuploidy. N Engl J Med. 2021 Nov 25;385(22):2047-2058. doi: 10.1056/NEJMoa2103613. PMID 34818479
- [Result] Smith ZD, Meissner A. DNA methylation: roles in mammalian development. Nat Rev Genet. 2013 Mar;14(3):204-20. doi: 10.1038/nrg3354. Epub 2013 Feb 12. PMID 23400093
- [Result] Jones PA. Functions of DNA methylation: islands, start sites, gene bodies and beyond. Nat Rev Genet. 2012 May 29;13(7):484-92. doi: 10.1038/nrg3230. PMID 22641018
- [Result] Jiang L, Zhang J, Wang JJ, Wang L, Zhang L, Li G, Yang X, Ma X, Sun X, Cai J, Zhang J, Huang X, Yu M, Wang X, Liu F, Wu CI, He C, Zhang B, Ci W, Liu J. Sperm, but not oocyte, DNA methylome is inherited by zebrafish early embryos. Cell. 2013 May 9;153(4):773-84. doi: 10.1016/j.cell.2013.04.041. PMID 23663777
- [Result] Li G, Yu Y, Fan Y, Li C, Xu X, Duan J, Li R, Kang X, Ma X, Chen X, Ke Y, Yan J, Lian Y, Liu P, Zhao Y, Zhao H, Chen Y, Sun X, Liu J, Qiao J, Liu J. Genome wide abnormal DNA methylome of human blastocyst in assisted reproductive technology. J Genet Genomics. 2017 Oct 20;44(10):475-481. doi: 10.1016/j.jgg.2017.09.001. Epub 2017 Sep 6. PMID 29037989
- [Result] Hardarson T, Van Landuyt L, Jones G. The blastocyst. Hum Reprod. 2012 Aug;27 Suppl 1:i72-91. doi: 10.1093/humrep/des230. Epub 2012 Jul 3. No abstract available. PMID 22763375
- [Result] Schieve LA, Meikle SF, Peterson HB, Jeng G, Burnett NM, Wilcox LS. Does assisted hatching pose a risk for monozygotic twinning in pregnancies conceived through in vitro fertilization? Fertil Steril. 2000 Aug;74(2):288-94. doi: 10.1016/s0015-0282(00)00602-6. PMID 10927046
- [Result] Fiorentino F, Biricik A, Bono S, Spizzichino L, Cotroneo E, Cottone G, Kokocinski F, Michel CE. Development and validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of embryos. Fertil Steril. 2014 May;101(5):1375-82. doi: 10.1016/j.fertnstert.2014.01.051. Epub 2014 Mar 6. PMID 24613537